CLINICAL TRIAL: NCT01718652
Title: An Open-Label, Single Sequence Study to Assess the Effect of a Single Dose of Cyclosporine on the Steady-State Pharmacokinetics of JNJ-28431754 (Canagliflozin) in Healthy Adult Subjects
Brief Title: A Study to Assess the Effects of Cyclosporine on the Pharmacokinetics and Safety of Canagliflozin (JNJ-28431754) in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR017926; 28431754DIA1031 (Other: Johnson & Johnson Pharmaceutical Research & Development, L.L.C); 2010-021854-21 (EudraCT Number)
Record Dates: First submitted 2012-10-29; First posted 2012-10-31 (Estimated); Last update posted 2012-11-27 (Estimated); Status verified 2012-11

CONDITIONS: Healthy
Keywords: Healthy; Canagliflozin (JNJ-28431754); Pharmacokinetics; Cyclosporine
MeSH Terms: interventions — Canagliflozin; Cyclosporine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Canagliflozin + cyclosporine (Experimental): Each volunteer will receive canagliflozin (JNJ-28431754) once daily on Days 1 through 8 with a single dose of cyclosporine on Day 7.
  Interventions: Drug: Canagliflozin (JNJ-28431754); Drug: Cyclosporine

INTERVENTIONS:
Drug: Canagliflozin (JNJ-28431754) — One 300 mg capsule-shaped tablet taken orally (by mouth) on Days 1 through 8.
  Other Names: JNJ-28431754
Drug: Cyclosporine — Four 100 mg capsules (400 mg total dose) taken orally 30 minutes before the last dose of canagliflozin (JNJ-28431754) on Day 8.

SUMMARY:
The purpose of this study is to determine how a single dose of cyclosporin affects the pharmacokinetics (ie, how the body affects the drug) of multiple doses of canagliflozin (JNJ-28431754). The safety and tolerability of canagliflozin will also be assessed in healthy volunteers.

DETAILED DESCRIPTION:
This study will be an open label (all volunteers and study staff know the identity of assigned treatments), single-center, multiple-dose study to determine how cyclosporin (a drug which reduces the activity of a patient's immune system) affects the pharmacokinetics of canagliflozin (a drug currently being investigated for the treatment of type 2 diabetes mellitus). The study will consist of 3 phases: a screening phase, an open-label treatment phase, and an end-of study (or follow-up) phase. Each volunteer will participate in the study for approximately 47 days.

ELIGIBILITY:
Inclusion Criteria:

* Must have body mass index between 18 and 30 kg/m2 (inclusive), and body weight not less than 50 kg
* If a woman, must be either postmenopausal, defined as no spontaneous menses for at least 18 months or amenorrhea for at least 6 months or surgically sterile (have had a hysterectomy, or tubal ligation)

Exclusion Criteria:

* History of smoking or use of nicotine-containing substances within the previous 2 months
* Have had history of or current medical illness considered to be clinically significant by the Investigator

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2011-02; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Plasma concentrations of canagliflozin (JNJ-28431754) | Day 7 and Day 8
  Comparison of the maximum plasma concentration (Cmax) and the area under the plasma concentration-time curve (AUC) of canagliflozin (JNJ-28431754) (measures of the body's exposure to canagliflozin) before and after administration of a single dose of cyclosporine. This will be used to determine whether there is a pharmacokinetic interaction between cyclosporine and canagliflozin.

SECONDARY OUTCOMES:
The number of volunteers with adverse events as a measure of safety and tolerability | Up to 47 days

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development,L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.
Locations (1):
- Antwerp, Belgium